CLINICAL TRIAL: NCT04506775
Title: Comparison of a Standalone, Continuous, Non-invasive Blood Pressure Monitor (cNIBP) to Radial Arterial Catheterization in Patients Undergoing Surgery.
Brief Title: Comparison of Non-invasive and Invasive Blood Pressure Monitors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Massachusetts, Worcester (Other)
Collaborators: Dynocardia, Inc (Industry)
Responsible Party: Principal Investigator, James Aaron Scott, Assistant Professor of Anesthesiology & Perioperative Medicine, University of Massachusetts, Worcester
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: H00019883
Record Dates: First submitted 2020-07-13; First posted 2020-08-10 (Actual); Results first posted 2025-09-10 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-08

CONDITIONS: Blood Pressure; Surgery; Intensive Care Unit
Keywords: Blood Pressure; BP; Surgery; Radial Artery Catheter

STUDY DESIGN:
Intervention Model Description: Single group design, patients are their own control.
Masking Description: None, patients are their own control.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Wrist one (Experimental): Wrist one will have both the ViTrack wrist cuff on one wrist
  Interventions: Device: ViTrack
- Wrist Two (Active Comparator): Wrist two and the radial artery catheter in the opposite wrist.
  Interventions: Procedure: Radial artery catheterization

INTERVENTIONS:
Device: ViTrack — ViTrack is a continuous non-invasive wearable blood pressure cuff.
  Arms: Wrist one
Procedure: Radial artery catheterization — Radial artery catheterization is the standard of care for measuring blood pressure continuously throughout surgery.
  Arms: Wrist Two

SUMMARY:
To compare a noninvasive and continuous radial artery blood pressure measurements utilizing ViTrack (developed by Dynocardia) to the standard of care radial artery catheterization, in patients undergoing surgery or those who are being cared for in the intensive care unit

DETAILED DESCRIPTION:
The ViTrack is strapped over the radial artery at the wrist.The ViTrack blood pressure cuff will be utilized to obtain continuous blood pressure (BP) readings throughout the surgical procedure or intensive care unit. This will allow us to compare BP readings between the non-invasive ViTrack device and the standard of care invasive intra-arterial catheters readings. Data collection from both the ViTrack and arterial catheter occur in the opposite wrists.

ELIGIBILITY:
Inclusion Criteria:

* Patients between the ages of 18 - 90 years age who are undergoing any surgery or in the intensive care unit and require intra-arterial catheterization for continuous BP measurement.
* Patients having elective surgeries.
* Patients having emergent surgeries, but only if research staff can have appropriate time to review study with patient and obtain signature on fact sheet prior to administration of medications that could affect coherency.
* Patients who are able to review, verbalize understanding, and sign fact sheet. If patient has a health care proxy (HCP) or legal guardian, study will be reviewed, and signature of HCP or legal guardian will be obtained.

Exclusion Criteria:

* Inability to obtain consent from the patient, HCP or legal guardian
* Greater than 10% difference in BP measurements between both arms prior to surgery
* Pregnant women
* Prisoners
* Inability to insert a radial artery catheter
* Any other condition that would increase the risk of participation in the study in the opinion of the site Investigator
* Upper extremity arteriovenous haemodialysis shunt
* Upper extremity amputation
* Surgical position/draping precludes access to the wrist.
* Wrist distortion or pain from arthritis
* Prior trauma or surgery at the radial artery monitoring site

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2024-04-18 (Actual); Study Completion 2024-04-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James A Scott, DO, Principal Investigator — University of Massachusetts, Worcester
Locations (1):
- University of Massachusetts Medical School, Worcester, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
Results and de-identified data will be securely shared with the sponsor. Sponsor may only see subject initials and study ID #. All other data will de-identified for review purposes and transferred via a secure method following the universities data sharing agreement with the sponsor.
Supporting Information: Study Protocol, SAP
Time Frame: Data will become available following data analysis within 12 months of study completion and will remain available for up to 3 years.
Access Criteria: Data will be accessed via secure methods outlined in a data sharing agreement.

REFERENCES:
- [Result] Heard SO, Lisbon A, Toth I, Ramasubramanian R. An evaluation of a new continuous blood pressure monitoring system in critically ill patients. J Clin Anesth. 2000 Nov;12(7):509-18. doi: 10.1016/s0952-8180(00)00201-4. PMID 11137411

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Wrist
Groups:
- All Study Participants: Wrist one will have the ViTrack wrist cuff on one wrist. ViTrack: ViTrack is a continuous non-invasive wearable blood pressure cuff.
  Wrist two with the radial artery catheter in the opposite wrist. Radial artery catheterization: Radial artery catheterization is the standard of care for measuring blood pressure continuously throughout surgery.
Period: Overall Study
Arm/Group | All Study Participants
Started | 30; 30 Wrist
Wrist 1 (Control) | 30; 30 Wrist
Wrist 2 (ViTrack) | 30; 30 Wrist
Completed | 30; 30 Wrist
Not Completed | 0; 0 Wrist

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: Wrist one will have both the ViTrack wrist cuff on one wrist. ViTrack: ViTrack is a continuous non-invasive wearable blood pressure cuff.
  Wrist two and the radial artery catheter in the opposite wrist. Radial artery catheterization: Radial artery catheterization is the standard of care for measuring blood pressure continuously throughout surgery.
Arm/Group | All Study Participants
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 9
  >=65 years | 21
Age, Continuous [Mean (Full Range); unit: Years] | 69.4 [53 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 22
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 30

OUTCOME MEASURES:

1. Primary Outcome: Comparison of Diastolic Blood Pressure
Description: 255 time points compared across continuous blood pressure (mmHg)
  As per the FDA standard ANSI/AAMI SP10:2008 or the newly adopted ISO 81060-3:2022 standard, the mean error should be <5mmHg or <6mmHg and the standard deviation should be <8mmHg or <10mmHg respectively.
Time Frame: Up to 24 Hours
Population: Wrist 1, the ViTrack wrist cuff represents the experimental arm of the study. Wrist 2, the radial arterial catheter, represents the gold standard arterial blood pressure monitor that the ViTrack device is being compared to. The outcome DBP for the ViTrack device reports the mean error and standard deviation for the ViTrack device in comparison to the gold standard in alignment with the FDA standards.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | All Study Participants
Number analyzed (Participants) | 30
mmHg | 0.90 (5.97)
Statistical Analysis 1: Comparison: All Study Participants; Test type: Non-Inferiority — As per the FDA standard ANSI/AAMI SP10:2008 or the newly adopted ISO 81060-3:2022 standard, the mean error should be <5mmHg or <6mmHg and the standard deviation should be <8mmHg or <10mmHg respectively; As per the FDA standard ANSI/AAMI SP10:2008 or the newly adopted ISO 81060-3:2022 standard, the mean error should be <5mmHg or <6mmHg and the standard deviation should be <8mmHg or <10mmHg respectively; Mean Error = 0.90

2. Primary Outcome: Comparison of Systolic Blood Pressure
Description: as for outcome 1
Time Frame: Up to 24 Hours
Population: Wrist 1, the ViTrack wrist cuff represents the experimental arm of the study. Wrist 2, the radial arterial catheter, represents the gold standard arterial blood pressure monitor that the ViTrack device is being compared to. The outcome SBP for the ViTrack device reports the mean error and standard deviation for the ViTrack device in comparison to the gold standard in alignment with the FDA standards.
Measure: Mean (Standard Deviation); unit: mmHg
Groups:
- All Study Participants: Wrist one will have both the ViTrack wrist cuff on one wrist ViTrack: ViTrack is a continuous non-invasive wearable blood pressure cuff.
  Wrist two and the radial artery catheter in the opposite wrist. Radial artery catheterization: Radial artery catheterization is the standard of care for measuring blood pressure continuously throughout surgery.
Arm/Group | All Study Participants
Number analyzed (Participants) | 30
mmHg | 0.19 (5.70)
Statistical Analysis 1: Comparison: All Study Participants; Test type: Non-Inferiority — As per the FDA standard ANSI/AAMI SP10:2008 or the newly adopted ISO 81060-3:2022 standard, the mean error should be < 5mmHg or <6mmHg and the standard deviation should be <8mmHg or <10mmHg respectively; As per the FDA standard ANSI/AAMI SP10:2008 or the newly adopted ISO 81060-3:2022 standard, the mean error should be < 5mmHg or <6mmHg and the standard deviation should be <8mmHg or <10mmHg respectively; Mean Error = 0.19 — As per the FDA standard ANSI/AAMI SP10:2008 or the newly adopted ISO 81060-3:2022 standard, the mean error should be < 5mmHg or <6mmHg and the standard deviation should be <8mmHg or <10mmHg respectively; As per the FDA standard ANSI/AAMI SP10:2008 or the newly adopted ISO 81060-3:2022 standard, the mean error should be < 5mmHg or <6mmHg and the standard deviation should be <8mmHg or <10mmHg respectively

3. Secondary Outcome: Skin Irritation
Description: Examining for local skin irritation
Time Frame: Up to 72 hours
Measure: Count of Participants; unit: Participants
Arm/Group | All Study Participants
Number analyzed (Participants) | 30
Participants | 0

ADVERSE EVENTS:
Time Frame: Date of enrollment only
Description: This device is non-invasive and has no inherent risk of serious adverse events or all-cause mortality
Arm/Group | All Study Participants
All-Cause Mortality (participants affected / at risk) | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2023-07-03): https://cdn.clinicaltrials.gov/large-docs/75/NCT04506775/Prot_001.pdf
  • Statistical Analysis Plan (2023-07-03): https://cdn.clinicaltrials.gov/large-docs/75/NCT04506775/SAP_002.pdf